CLINICAL TRIAL: NCT00923364
Title: Pilot and Feasibility Study of Reduced-Intensity Hematopoietic Stem Cell Transplant for Patients With GATA2 Mutations
Brief Title: Pilot and Feasibility Study of Reduced-Intensity Hematopoietic Stem Cell Transplant for MonoMAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dennis Hickstein, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090096; 09-C-0096; NCT00884923 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: MDS; Immunodeficiency; GATA2
Keywords: GATA2; Transplant; Immunodeficiency; Myelodysplasia; MonoMAC
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Anemia, Refractory, with Excess of Blasts; GATA2 Deficiency | interventions — Cyclophosphamide; fludarabine phosphate; Whole-Body Irradiation; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Recipients and Healthy Related Donors (Experimental): Hematopoietic Stem Cell Transplant for MonoMAC: 10/10 Human Leukocyte Antigen (HLA) Matched Related Donor (MRD) or Unrelated Donor (URD) Transplant. 9/10 HLA Matched Related Donor or Unrelated Donor Transplant. Haploidentical Related Donor Transplant. Umbilical Cord Blood Transplant.
  Interventions: Drug: Cyclophosphamide (CTX, Cytoxan); Drug: Fludarabine(Fludara,Berlex Laboratories); Procedure: Total Body Irradiation (TBI); Procedure: Allogeneic Hematopoietic Stem Cell (HSC); Drug: Equine Anti-Thymocyte Globulin

INTERVENTIONS:
Drug: Cyclophosphamide (CTX, Cytoxan) — 14.5 mg/kg intravenous (IV) (in the vein) infusion over 30 minutes once daily on days -6 and -5 (weight based dosing) or 50 mg/kg IV infusion over 2 hours on day -6 (weight based dosing) or 50/kg IV once daily x 2 doses on days +3 and +4
  Other Names: Cytoxan
Drug: Fludarabine(Fludara,Berlex Laboratories) — 40 mg/m2 IV (in the vein) over 30 minutes (in the vein) once daily on Days -6, -5, -4, and -3 or 30 mg/m(2) IV over 30 minutes (in the vein) once daily on Days -6, -5, -4, -3, and -2
  Other Names: Fludara
Procedure: Total Body Irradiation (TBI) — 200 centigray (cGy) on Day -1 or 300 cGy on Day -1 (for 9/10 URD and Haplo patients)
  Other Names: TBI
Procedure: Allogeneic Hematopoietic Stem Cell (HSC) — stem cell transplant
Drug: Equine Anti-Thymocyte Globulin — 30mg/kg IV (in the vein) once daily x 3 days on Days -6, -5, -4 (3 doses total)
  Other Names: ATG

SUMMARY:
Background:

* Stem cells are immature blood cells that grow in the bone marrow and produce all of the cells needed for normal blood and immunity. Stem cells can be taken from one person (donor) and given to another person (recipient) through allogeneic stem cell transplantation. Donor stem cells can then replace the recipients stem cells in the bone marrow, restoring normal blood production and immunity. Most allogeneic transplants now use stem cells collected from the donors blood in a process called peripheral blood stem cell transplantation.
* Monocytopenia and mycobacterial infection (MonoMAC) is an immunodeficiency disease that is characterized by a lack of monocytes, a type of white blood cell, and an increased risk of developing mycobacteria infections that may cause tuberculosis.
* Allogeneic stem cell transplantation has been used successfully to treat many kinds of immune diseases and cancers that develop in blood or immune system cells. Researchers have been studying a particular kind of stem cell transplantation that uses lower than usual doses of chemotherapy and particular combinations of drugs to improve the results of the procedure for patients with blood-related cancers and pre-cancerous conditions.

Objectives:

* To determine the safety and efficacy of reduced-intensity hematopoietic stem cell transplants (a particular stem cell transplantation procedure) for treating MonoMAC.

Eligibility:

* Patients 18-60 years of age who have MonoMAC and who have been matched with a suitable stem cell donor.

Design:

* Donors and recipients will undergo separate procedures as part of this protocol.
* Donors:
* National Institutes of Health researchers will take the donor s medical history, perform a physical exam, take blood samples, and explain the procedure. Tests will be performed to check the donors heart, lung, kidney, and liver function.
* Donors will receive injections of a drug called filgrastim (G-CSF), which causes stem cells to travel from bone marrow into blood. The G-CSF shots will be given for 5 to 7 days before the collection procedure.
* Donors will undergo apheresis to collect white blood cells and stem cells directly from the blood, which can be done as an outpatient procedure. Researchers may consider the alternative of directly collecting bone marrow from the donor, which will require an overnight hospital stay.
* Recipients:
* Recipients will receive 3 days of pre-transplant chemotherapy and radiation therapy to prepare for the transplant. For 4 days before the transplant, recipients will receive the chemotherapy drug fludarabine, followed by a single dose of radiation therapy, and will also receive the drugs tacrolimus and sirolimus to prevent the donor cells from attacking the recipient s normal tissues.
* Recipients will then receive the transplant of donor stem cells and will continue to receive tacrolimus and sirolimus for 3 months after the transplant to prevent the donor cells from attacking the recipient s normal tissues. Recipients will be discharged from the hospital once their condition is stable.
* Recipients will visit the NCI clinic regularly for the first 5 months after the transplant, and then less often for at least 5 years. Recipients may receive additional donor immune cells (donor lymphocyte infusion) after the transplant if the study doctors believe they are needed.

DETAILED DESCRIPTION:
BACKGROUND:

Mutations in GATA binding protein 2 (GATA2) lead to an immunodeficiency disease that transforms into myelodysplastic syndrome (MDS) and acute myelogenous leukemia (AML). This syndrome, previously known as MonoMAC, has 4 clinical features: 1) infections with Mycobacterium Avium Complex (MAC) and other opportunistic infections as a teenager or young adult, 2) a peripheral blood leukocyte flow cytometry profile with T-lymphocytes, but a severe deficiency of monocytes, B-lymphocytes, and Natural Killer (NK) cells, 3) the propensity to progress to MDS/AML, and 4) mutations in the gene GATA2. In this pilot study we propose to evaluate the efficacy and safety of a reduced intensity allogeneic hematopoietic stem cell transplantation (HSCT) regimen for patients with mutations in GATA2. We are particularly interested in determining whether allogeneic HSCT using this regimen reconstitutes normal hematopoiesis in patients with mutations in GATA2.

OBJECTIVES:

Primary Objective:

* To determine efficacy, namely whether reduced-intensity allogeneic HSCT results in engraftment and restores normal hematopoiesis by day +100 in patients with mutations in GATA2.
* To determine the safety of this HSCT regimen in patients with mutations in GATA2, including transplant related toxicity, the incidence of acute and chronic graft-versus host disease, immune reconstitution, overall survival, and disease-free survival

ELIGIBILITY:

Eligibility includes patients 12-60 years old with mutations in GATA2 who have a life expectancy of > 3 months but < 24 months, and who have a 10/10 matched related donor, a 10/10 or 9/10 matched unrelated donor (HLA -A, -B, -C, DRB1, DQB1 by high resolution typing identified through the National Marrow Donor Program), a 4/6 (or greater human leukocyte antigens (HLA -A), -B, DRB1) matched unrelated umbilical cord donor, or a haploidentical donor. Patients with GATA2 mutations who are 12-17 years of age are required to have MDS with chromosomal abnormalities to be eligible for this protocol.

DESIGN:

* Patients with mutations in GATA2 with a 10/10 matched related or 10/10 matched unrelated donor, will receive a reduced-intensity pre-transplant conditioning regimen consisting of fludarabine 30 mg/m(2)/day on days -4, -3, and -2, 200 centigray (cGy) total body irradiation (TBI) on day -1, and HSCT on day 0. Patients with mutations in GATA2 and a 9/10 matched unrelated donor will receive a reduced-intensity pre-transplant conditioning regimen consisting of fludarabine 30 mg/m(2)/day on days -4, -3, and -2, 300cGy total body irradiation (TBI) on day -1, and HSCT on day 0. Patients with mutations in GATA2 with umbilical cord blood units will receive a reduced-intensity conditioning regimen with cyclophosphamide 50 mg/kg on day -6, fludarabine 40 mg/m(2) on days -6 to -2, equine anti-thymocyte globulin (ATG) 30 mg/kg intravenous (IV) on days -6, -5 and -4, 200 cGy TBI on day -1, and HSCT on day 0. Patients with a haploidentical donor will receive a reduced intensity-conditioning regimen with cyclophosphamide 14.5 mg/kg on days -6 and -5, fludarabine 30 mg/m(2) on 4days -6 to -2, and 200 cGy TBI on day -1. Donor bone marrow cells will be infused on day 0.
* Post-transplant immunosuppression for graft-versus-host-disease prophylaxis will consist of sirolimus (Rapamycin) and tacrolimus until day +180, provided that there is no evidence of graft-versus-host disease. Post-transplant immunosuppression for graft versus-host-disease prophylaxis for recipients of haploidentical donors will consist of cyclophosphamide 50 mg/kg on days +3 and +4, along with sirolimus from day +5 to day 180, and tacrolimus from day +5 to day 180, providing that there is no graft-versus-host disease (GVHD).

ELIGIBILITY:
* INCLUSION CRITERIA RECIPIENT:

  1. Patient age of 12-60 years
  2. GATA2 Mutation Syndrome

     1. Clinical history of at least two episodes of life-threatening infection with opportunistic organisms, one of which is a MAC infection.
     2. Mutation in the GATA2 gene performed by the CLIA certified laboratory of Dr. Steven Holland of the NIAID Institute of the NIH.
  3. Available 10/10 HLA-matched related or 8/8 matched unrelated donor, or 4/6 (or greater) matched UCB unit(s) with a total dose of greater than or equal to 3.5 times 10(7) TNC/kg.
  4. Patients may have evidence of MDS with one or more peripheral blood cytopenias and greater than 5% blasts but less than 10% blasts in the bone marrow in the absence of GCSF.

     Patients previously treated for acute myelogenous leukemia are eligible if they have less than or equal to 10% blasts in the bone marrow in the absence of G-CSF.

     Subjects 12-17 years of age are required to have MDS with chromosomal abnormalities in addition to mutation in the GATA2 gene for enrollment on this protocol.
  5. Left ventricular ejection fraction > 50%, preferably by 2-D echo, or by MUGA, or shortening fraction > 28% by ECHO, obtained within 28 days of enrollment.
  6. Pulmonary Function Tests: Adult patients: DLCO diffusion capacity and FEV1 greater than 10% of expected value obtained within 28 days of enrollment. Pediatric patients: DLCO corrected for hemoglobin and alveolar volume greater than or equal to 20% of predicted.
  7. Creatinine: Adult patients: less than or equal to 2.0 mg/dl and creatinine clearance greater than or equal to 30 ml/min; Pediatric patients: age-adjusted normal serum creatinine OR a creatinine clearance > 60 mL/min/1.73m(2).
  8. Serum total bilirubin less than 2.5 mg/dl; ALT and AST less than or equal to 5 times upper limit of normal .
  9. Adequate central venous access potential.
  10. Written informed consent/assent obtained from patient/parent or legal guardian.
  11. Life expectancy of at least 3 months but less than 24 months.
  12. Disease status: Patients are to be referred in remission for evaluation. Should a patient have progressive disease or a donor not be available after enrollment, the patient will be referred back to their primary hematologist-oncologist for treatment. If this course of action is not in the best interest of the patient according to the clinical judgment of the PI/LAI, then the patient may receive standard treatment for the malignant disease under the current study. If under either of these settings, it becomes apparent that the patient will not be able to proceed to transplant, then he/she must come off study. Recipient-Subjects receiving a standard therapy will be told about the therapy, associated risks, benefits alternatives of the proposed therapy, and availability of receiving the same treatment elsewhere, outside of a research protocol.

EXCLUSION CRITERIA- RECIPIENT:

1. HIV infection.
2. Chronic active hepatitis B. Patient may be hepatitis B core antibody positive. For patients with a concomitant positive hepatitis B surface antigen, patients will require a hepatology consultation. The risk-benefit profile of transplant and hepatitis B will be discussed with the patient, and eligibility determined by the PI and the protocol chairperson.
3. History of psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent.
4. Active infection that is not responding to antimicrobial therapy.
5. Active CNS involvement by malignancy (patients with known positive CSF cytology or parenchymal lesions visible by CT or MRI.
6. Pregnant or lactating.
7. Sexually active individuals capable of becoming pregnant who are unable or unwilling to use effective form(s) of contraception during time enrolled on study and for 1 year post-transplant. Effective forms of contraception include one or more of the following: intrauterine device (IUD), hormonal (birth control pills, injections, or implants), tubal ligation/hysterectomy, partners vasectomy, barrier methods, (condom, diaphragm, or cervical cap), or abstinence. The effects on breast-milk are also unknown and may be harmful to the infant; therefore, women should not breast feed during the interval from study entry to one year post-transplant. Males on the protocol must use an effective form of contraception at study entry, and for one year post-transplant. The effects of transplant, the radiation, and the medications used after transplant may be harmful to a fetus.
8. Presence of active malignancy in another organ system other than the hematopoietic
9. No available 10/10 HLA-matched related or 8/8 matched unrelated donor, or 4/6 (or greater) matched UCB unit(s) with a total dose of greater than or equal to 3.5 times 10(7) TNC/kg.
10. Lack of mutation in GATA2 as demonstrated by the CLIA certified laboratory of Dr. Steven Holland in the NIAID.

INCLUSION CRITERIA- MATCHED RELATED DONOR:

1. Related donor matched at HLA-A, B, C, DR, and DQ loci by high resolution typing (10/10 antigen/allele match) are acceptable donors.
2. Matched related donors for pediatric recipients must be 18 years of age or older. If more than one matched related donor is available, we will select the oldest donor to further decrease the risk of potential disease transmission.
3. Ability to give informed consent.
4. Age 18-60 years.
5. No history of life-threatening opportunistic infection.
6. Adequate venous access for peripheral apheresis, or consent to use a temporary central venous catheter for apheresis.
7. Donors must be HIV negative, hepatitis B surface antigen negative, and hepatitis C antibody negative. This is to prevent the possible transmission of these infections to the recipient.
8. A donor who is lactating must be willing and able to interrupt breast-feeding or substitute formula feeding for her infant during the period of filgrastim administration and for two days following the final dose. Filgrastim may be secreted in human milk, although its bioavailability from this source is not known. Limited clinical data suggest that short-term administration of filgrastim or sargramostim to neonates is not associated with adverse outcomes.

INCLUSION CRITERIA- MATCHED UNRELATED DONOR:

1. Unrelated donor matched at 10/10 or 9/10 HLA-A, B, C, DRB1, and DQB1 loci by high resolution typing.
2. Matched unrelated donors for pediatric recipients must be 18 years of age or older.
3. The evaluation of donors shall be in accordance with existing NMDP Standard Policies and Procedures. General donor inclusion criteria specified in the NMDP Standard.

EXCLUSION CRITERIA- MATCHED RELATED DONOR:

1. Age less than 18 years.
2. HIV infection.
3. Chronic active hepatitis B. Donor may be hepatitis core antibody positive.
4. History of psychiatric disorder which in the opinion of the PI may compromise compliance with transplant protocol, or which does not allow to be appropriately informed.
5. History of hypertension that is not controlled by medication, stroke, or severe heart disease. Individuals with symptomatic angina will be considered to have severe heart disease and will not be eligible to be a donor.
6. Other medical contraindications to stem cell donation (i.e. severe atherosclerosis, autoimmune disease, iritis or episcleritis, deep venous thrombosis, cerebrovascular accident).
7. History of prior malignancy. However, cancer survivors who have undergone potentially curative therapy may be considered for stem cell donation on a case-by-case basis. The risk/benefit of the transplant and the possibility of transmitting viable tumor cells at the time of transplantation will be discussed with the patient.
8. Donors must not be pregnant. Pregnancy is an absolute contraindication under this protocol. The effects of cytokine administration on a fetus are unknown. Donors of childbearing potential must use an effective method of contraception. Effective forms of contraception include one or more of the following: intrauterine device (IUD), hormonal (birth control pills, injections, or implants), tubal ligation/hysterectomy, partner s vasectomy, barrier methods, (condom, diaphragm, or cervical cap), or abstinence.
9. Thrombocytopenia (platelets less than 150,000 per micro l) at baseline evaluation.
10. Donors receiving experimental therapy or investigational agents.
11. Sensitivity to filgrastim or to E. coli-derived recombinant protein products.
12. History of autoimmune disorders, with the exception of thyroid disorders.
13. History of documented deep vein thrombosis or pulmonary embolism.

EXCLUSION CRITERIA- MATCHED UNRELATED DONOR:

Failure to qualify as an NMDP donor

INCLUSION CRITERIA- UMBILICAL CORD BLOOD UNIT-HLA TYPING AND DOSE

1. At least an HLA UCB 4/6 match (Class I-A, B by low resolution, and Class II-DR by high resolution) to recipient. The following algorithm will be applied to determine if patient will receive single or double umbilical cord graft:
2. For Single UCB SCT:

   * If 6/6 match the unit must have > 3 x 10(7) nucleated cells /kg of recipient body weight.
   * If 5/6 match the unit must have > 4 x 10(7) nucleated cells /kg of recipient body weight.
   * If 4/6 match the unit must have > 5 x 10(7) nucleated cells/kg of recipient body weight. Recipient body weight will be determined as per standard guidelines.
3. If no single UCB with the above characteristics is available, a double UCB will be considered. Units will be selected with the following criteria:

   * Both units will be at least 4/6 match (Class I-A, B by low resolution, Class II-DR by high resolution) to recipient, and should be at least a 4/6 match (Class I-A, B by low resolution, Class II-DR by high resolution) to each other.
   * At least one UCB will have a minimum cell dose of 2.0 X 10(7) TNC/kg of recipient body weight.
   * The minimum combined dose of both units must be at least 3.5 x 10(7) TNC/kg of recipient body weight.
   * The smaller of the two units (UCB2) will have a minimum of 1.5 X 10(7) TNC/kg of recipient body weight.
   * The TNC of non-RBC reduced units will be dose corrected by -25% to allow for cell loss while washing the unit.

INCLUSION CRITERIA- HAPLOIDENTICAL RELATED DONOR:

* A haploidentical donor that shares one haplotype in common with the recipient such that HLA compatibility will be a minimum of 5 out of 10 HLA loci matched. The HLA loci to be tested will be HLA A, B, Cw, DRB1, and DQB1. A minimum number of mismatches is desirable; however if several options are available the selection of a donor will be based on the loci where the mismatch occurs and the relative importance of its potential immunological function. Donor-recipient pairs will initially be typed molecularly to provide a low resolution typing (antigen-level) to aid in the selection of the potential donor. Upon review of the familial inheritance pattern, a qualified HLA staff member will review haplotype inheritance. High resolution (allele-level) typing will be performed. Final selection of a donor will be in consultation with NCI physicians and qualified HLA personnel. Haploidentical related donors for pediatric recipients must be 15 years of age or older. If more than one haploidentical related donor is available, we will evaluate each donor individually according to overall health, ABO matching, cytomegalovirus (CMV), etc. to select the donor
* Age 15-60 years
* No history of life-threatening opportunistic infection
* Adequate venous access for peripheral apheresis, or consent to use a temporary central venous catheter for apheresis.
* Donors must be HIV negative, hepatitis B surface antigen negative, and hepatitis C antibody negative. This is to prevent the possible transmission of these infections to the recipient.
* Haploidentical donors will undergo marrow harvest with general anesthesia. Subjects will undergo anesthesia consultation, and meet criteria for eligibility/enrollment. CD34+ fraction will be determined.
* Subjects will also undergo the Donor Health History Screen to determine donor eligibility using standard DTM criteria in the Dowling Apheresis Clinic by skilled staff in the Blood Services Section for adult patients and age-appropriate questioning when indicated for pediatric subjects.
* Subjects will undergo follow-up history and physical examination within 1 week of donation.

EXCLUSION CRITERIA- HAPLOIDENTICAL DONOR:

* Age less than 15 years.
* HIV infection
* Chronic active hepatitis B. Donor may be hepatitis core antibody positive.
* History of psychiatric disorder which in the opinion of the PI may compromise compliance with transplant protocol, or which does not allow for appropriate informed
* History of hypertension that is not controlled by medication, stroke, or severe heart disease. Individuals with symptomatic angina will be considered to have severe heart disease and will not be eligible to be a donor.
* Other medical contraindications to stem cell donation (i.e. severe atherosclerosis, autoimmune disease, iritis or episcleritis, deep venous thrombosis, cerebrovascular accident)
* History of prior malignancy. However, cancer survivors who have undergone potentially curative therapy may be considered for stem cell donation on a case-by-case basis. The risk/benefit of the transplant and the possibility of transmitting viable tumor cells at the time of transplantation will be discussed with the patient.
* Donors must not be pregnant. Pregnancy is an absolute contraindication under this protocol. The effects of cytokine administration on a fetus are unknown. Donors of childbearing potential must use an effective method of contraception. Effective forms of contraception include one or more of the following: intrauterine device (IUD), hormonal (birth control pills, injections, or implants), tubal ligation/hysterectomy, partners vasectomy, barrier methods, (condom, diaphragm, or cervical cap), or abstinence.
* Thrombocytopenia (platelets less than 150,000 per microliter) at baseline evaluation.
* Donors receiving experimental therapy or investigational agents.
* Sensitivity to filgrastim or to E. coli-derived recombinant protein products.
* History of autoimmune disorders, with the exception of thyroid disorders
* History of documented deep vein thrombosis or pulmonary embolism
* Mutation in GATA2

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2009-05-07 (Actual); Primary Completion 2014-06-12 (Actual); Study Completion 2017-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis D Hickstein, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anasetti C, Beatty PG, Storb R, Martin PJ, Mori M, Sanders JE, Thomas ED, Hansen JA. Effect of HLA incompatibility on graft-versus-host disease, relapse, and survival after marrow transplantation for patients with leukemia or lymphoma. Hum Immunol. 1990 Oct;29(2):79-91. doi: 10.1016/0198-8859(90)90071-v. PMID 2249952
- [Background] Anderlini P, Korbling M, Dale D, Gratwohl A, Schmitz N, Stroncek D, Howe C, Leitman S, Horowitz M, Gluckman E, Rowley S, Przepiorka D, Champlin R. Allogeneic blood stem cell transplantation: considerations for donors. Blood. 1997 Aug 1;90(3):903-8. PMID 9242518
- [Background] Antin JH, Kim HT, Cutler C, Ho VT, Lee SJ, Miklos DB, Hochberg EP, Wu CJ, Alyea EP, Soiffer RJ. Sirolimus, tacrolimus, and low-dose methotrexate for graft-versus-host disease prophylaxis in mismatched related donor or unrelated donor transplantation. Blood. 2003 Sep 1;102(5):1601-5. doi: 10.1182/blood-2003-02-0489. Epub 2003 May 1. PMID 12730113
- [Result] Cuellar-Rodriguez J, Gea-Banacloche J, Freeman AF, Hsu AP, Zerbe CS, Calvo KR, Wilder J, Kurlander R, Olivier KN, Holland SM, Hickstein DD. Successful allogeneic hematopoietic stem cell transplantation for GATA2 deficiency. Blood. 2011 Sep 29;118(13):3715-20. doi: 10.1182/blood-2011-06-365049. Epub 2011 Aug 3. PMID 21816832
- [Derived] West RR, Hsu AP, Holland SM, Cuellar-Rodriguez J, Hickstein DD. Acquired ASXL1 mutations are common in patients with inherited GATA2 mutations and correlate with myeloid transformation. Haematologica. 2014 Feb;99(2):276-81. doi: 10.3324/haematol.2013.090217. Epub 2013 Sep 27. PMID 24077845
- [Derived] Purisch SE, Shanis D, Zerbe C, Merideth M, Cuellar-Rodriguez J, Stratton P. Management of uterine bleeding during hematopoietic stem cell transplantation. Obstet Gynecol. 2013 Feb;121(2 Pt 2 Suppl 1):424-7. doi: 10.1097/aog.0b013e318270ecd3. PMID 23344397
- [Derived] Calvo KR, Vinh DC, Maric I, Wang W, Noel P, Stetler-Stevenson M, Arthur DC, Raffeld M, Dutra A, Pak E, Myung K, Hsu AP, Hickstein DD, Pittaluga S, Holland SM. Myelodysplasia in autosomal dominant and sporadic monocytopenia immunodeficiency syndrome: diagnostic features and clinical implications. Haematologica. 2011 Aug;96(8):1221-5. doi: 10.3324/haematol.2011.041152. Epub 2011 Apr 20. PMID 21508125
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0096.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Recipients: Hematopoietic Stem Cell Transplant for MonoMAC: 10/10 Human Leukocyte Antigen (HLA) Matched Related Donor (MRD) or Unrelated Donor (URD) Transplant. 9/10 HLA Matched Related Donor or Unrelated Donor Transplant. Haploidentical Related Donor Transplant. Umbilical Cord Blood Transplant.
  Fludarabine(Fludara,Berlex Laboratories): 40 mg/m(2) intravenous (IV) (in the vein) over 30 minutes (in the vein) once daily on Days -6, -5, -4, and -3 or 30 mg/m(2) IV over 30 minutes (in the vein) once daily on Days -6, -5, -4, -3, and -2
  Total Body Irradiation (TBI): 200 centigray (cGy) on Day -1 or 300 cGy on Day -1 (for 9/10 URD and Haplo patients)
  Allogeneic hematopoietic stem cell (HSC): stem cell transplant
Period: Overall Study
Arm/Group | Recipients | Healthy Related Donors
Started | 14 | 5
Completed | 10 | 5
Not Completed | 4 | 0
Not completed — Death | 3 | 0
Not completed — Did not go to transplant | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data were not collected separately for donors and recipients.
Groups:
- Recipients and Healthy Related Donors: Hematopoietic Stem Cell Transplant for MonoMAC: 10/10 Human Leukocyte Antigen (HLA) Matched Related Donor (MRD) or Unrelated Donor (URD) Transplant. 9/10 HLA Matched Related Donor or Unrelated Donor Transplant. Haploidentical Related Donor Transplant. Umbilical Cord Blood Transplant.
  Fludarabine(Fludara,Berlex Laboratories): 40 mg/m(2) intravenous (IV) (in the vein) over 30 minutes (in the vein) once daily on Days -6, -5, -4, and -3 or 30 mg/m(2) IV over 30 minutes (in the vein) once daily on Days -6, -5, -4, -3, and -2
  Total Body Irradiation (TBI): 200 centigray (cGy) on Day -1 or 300 cGy on Day -1 (for 9/10 URD and Haplo patients)
  Allogeneic hematopoietic stem cell (HSC): stem cell transplant Healthy related donors =5; recipients = 14.
Arm/Group | Recipients and Healthy Related Donors
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.21 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Days to Neutrophil Engraftment
Description: Neutrophil engraftment is defined as a neutrophil count of >0.5 x 10(9) cells/L for 3 consecutive days.
Time Frame: 30 days
Population: 10/19 analyzed:5 pts were healthy related donors, 1 pt taken off study prior to transplant & 3 pts had early deaths (before outcome measurements could be evaluated)
Measure: Median (Full Range); unit: Days
Groups:
- Recipients Only: Hematopoietic Stem Cell Transplant for MonoMAC: 10/10 Human Leukocyte Antigen (HLA) Matched Related Donor (MRD) or Unrelated Donor (URD) Transplant. 9/10 HLA Matched Related Donor or Unrelated Donor Transplant. Haploidentical Related Donor Transplant. Umbilical Cord Blood Transplant.
  Fludarabine(Fludara,Berlex Laboratories): 40 mg/m(2) intravenous (IV) (in the vein) over 30 minutes (in the vein) once daily on Days -6, -5, -4, and -3 or 30 mg/m(2) IV over 30 minutes (in the vein) once daily on Days -6, -5, -4, -3, and -2 Total Body Irradiation (TBI): 200 centigray (cGy) on Day -1 or 300 cGy on Day -1 (for 9/10 URD and Haplo patients) Allogeneic hematopoietic stem cell (HSC): stem cell transplant
Arm/Group | Recipients Only
Number analyzed (Participants) | 10
Days | 12 [12 to 80]

2. Primary Outcome: Days to Platelet Engraftment
Description: Platelet engraftment is defined as a platelet count of >20 x 10(9) cells/L for 7 consecutive days without requiring a platelet transfusion.
Time Frame: 30 days
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Recipients Only
Number analyzed (Participants) | 10
Days | 30 [0 to 30]

3. Secondary Outcome: Percentage of Donor Cells at Last Follow Up in Patients With Mutations GATA Binding Protein 2 (GATA2)
Description: Engraftment of donor cells was assessed using polymorphisms in regions known to contain short tandem repeats. Peripheral blood cluster of differentiation 14 (CD14+), cluster of differentiation 3 (CD3-)/cluster of differentiation 56 (CD56+), cluster of differentiation 19 (CD19+), and CD3+ subsets were isolated by flow cytometry and chimerism was assessed.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Full Range); unit: percentage of donor cells
Arm/Group | Recipients Only
Number analyzed (Participants) | 10
percentage of donor cells
  Donor CD14+ cells, % | 99.8 [99 to 100]
  Donor CD19+ cells, % | 100 [100 to 100]
  Donor CD3-/CD56+ cells, % | 99.8 [99 to 100]
  Donor CD3+ cells, % | 97.6 [91 to 100]

4. Secondary Outcome: Incidence of Acute and Chronic Graft-versus-host Disease (GVHD)
Description: Acute GVHD is assessed according to the 1994 Consensus Conference Grading Criteria. Chronic GVHD is assessed by the 2005 Chronic GVHD Consensus Project. GVHD can affect performance status and attack multiple organ systems such as the skin, liver, gut, mouth, eyes, joints, lung, etc. that can lead to a rash, diarrhea, metabolic changes, infection and/or death. The clinical grading of acute GVHD is grade 0 (none) to 4 (severe). Chronic GVHD is a delayed form of GVHD that may occur after day 100 post transplant.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Recipients Only
Number analyzed (Participants) | 10
participants
  Acute | 2
  Chronic | 3

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as date of on-study to date of death from any cause or last follow up.
Time Frame: 2 years
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Recipients Only
Number analyzed (Participants) | 10
months | 76 [18 to 95]

6. Secondary Outcome: Number of Participants With Disease Free Survival
Description: Number of participants with documented evidence of disease progression following start of treatment.
Time Frame: 2 years
Population: 10/19 analyzed:5pts were healthy related donors, 1 pt taken off study prior to transplant & 3 pts had early deaths (before outcome measurements could be evaluated)
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients Only
Number analyzed (Participants) | 10
Participants | 8

7. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events v3.0. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately, 91 months
Population: Data were not collected separately for donors and recipients.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipients and Healthy Related Donors
Number analyzed (Participants) | 19
Participants | 16

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately, 91 months.
Description: Data were not collected separately for donors and recipients.
Arm/Group | Recipients and Healthy Related Donors
All-Cause Mortality (participants affected / at risk) | 4/19
Serious Adverse Events (participants affected / at risk) | 12/19
Other Adverse Events (participants affected / at risk) | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipients and Healthy Related Donors (N=19)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (3)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac troponin I (cTnI) (Cardiac disorders) | 1 (1)
Cardiopulmonary arrest, cause unknown (non-fatal) (Cardiac disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
DIC (disseminated intravascular coagulation) (Vascular disorders) | 1 (1)
Death not associated with CTCAE term::Death NOS (General disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Febrile neutropenia (Infections and infestations) | 2 (4) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Hemorrhage, GI::Upper GI NOS (Gastrointestinal disorders) | 1 (2)
Hemorrhage, GU::Vagina (Renal and urinary disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory::Lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hepatobiliary/Pancreas - Other (Specify, __) (Hepatobiliary disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Gallbladder (cholecystitis)
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Sinus
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Urinary tract NOS
Infection - Other (Specify, __) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper aerodigestive NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 1 (1)
Infection with unknown ANC::Blood (Infections and infestations) | 1 (1)
Infection with unknown ANC::Colon (Infections and infestations) | 1 (1)
Leak (including anastomotic), GI::Leak NOS (Nervous system disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (3)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Mucositis/stomatitis (clinical exam)::Stomach (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (functional/symptomatic)::Esophagus (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
Pain::Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 2 (8)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Proteinuria (Metabolism and nutrition disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)
Vessel injury-artery::Other NOS (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recipients and Healthy Related Donors (N=19)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 2 (2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 11 (37)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 10 (38)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5 (20)
Alkaline phosphatase (Metabolism and nutrition disorders) | 6 (23)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ascites (non-malignant) (Gastrointestinal disorders) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 5 (12)
Bladder spasms (Renal and urinary disorders) | 1 (1)
CD4 count (Blood and lymphatic system disorders) | 1 (3)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1 (1)
Carbon monoxide diffusion capacity (DL(co)) (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Cardiac Arrhythmia - Other (Specify, persistent tachycardia) (Cardiac disorders) | 1 (1)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 2 (7)
Cystitis (Renal and urinary disorders) | 1 (1)
Dermal change lymphedema, phlebolymphedema (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatology/Skin - Other (Specify, v dermatitis per biopsy) (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (13)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 4 (4)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Edema: limb (Blood and lymphatic system disorders) | 2 (2)
Enteritis (inflammation of the small bowel) (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 3 (3)
FEV(1) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 3 (11) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 4 (8)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 4 (4)
Gastrointestinal - Other (Specify, v) (Gastrointestinal disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 3 (48)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 9 (72)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Metabolism and nutrition disorders) | 1 (1)
Hemorrhage, GI::Lower GI NOS (Gastrointestinal disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hemorrhage/Bleeding - Other (Specify, diathesis) (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (5)
Hypotension (Vascular disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Infection (documented clinically or microbiologically) (Infections and infestations) | 4 (9) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Catheter-related
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Pharynx
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Pleura (empyema)
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Rectum
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Spinal cord (myelitis)
Infection (documented clinically or microbiologically) (Infections and infestations) | 3 (4) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Urinary tract NOS
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Vagina
Infection (documented clinically or microbiologically) (Infections and infestations) | 2 (2) — with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Wound
Infection - Other (Specify, skin:zoster; thrush) (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Anal/perianal (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bladder (urinary) (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 9 (21)
Infection with normal ANC or Grade 1 or 2 neutrophils::Catheter-related (Infections and infestations) | 2 (5)
Infection with normal ANC or Grade 1 or 2 neutrophils::Ileum (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Larynx (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils::Nose (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Oral cavity-gums (gingivitis) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Peritoneal cavity (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Pharynx (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Sinus (Infections and infestations) | 3 (6)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper aerodigestive NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 3 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 3 (6)
Infection with normal ANC or Grade 1 or 2 neutrophils::Vulva (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Wound (Infections and infestations) | 1 (3)
Infection with unknown ANC::Blood (Infections and infestations) | 2 (5)
Infection with unknown ANC::Brain + Spinal cord (encephalomyelitis) (Infections and infestations) | 1 (1)
Infection with unknown ANC::Bronchus (Infections and infestations) | 1 (1)
Infection with unknown ANC::Catheter-related (Infections and infestations) | 1 (1)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with unknown ANC::Upper airway NOS (Infections and infestations) | 1 (1)
Leak, cerebrospinal fluid (CSF) (Nervous system disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 7 (90)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1)
Lymphedema-related fibrosis (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 9 (126)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 3 (9)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Mood alteration::Agitation (Nervous system disorders) | 1 (1)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 2 (3)
Muscle weakness, generalized or specific area (not due to neuropathy)::Facial (Musculoskeletal and connective tissue disorders) | 1 (2)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (7)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6 (20)
Ocular surface disease (Eye disorders) | 1 (1)
Ocular/Visual - Other (Specify, decreased vision) (Eye disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 4 (6)
Pain::Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Pain::Anus (Gastrointestinal disorders) | 1 (1)
Pain::Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 2 (4)
Pain::Dental/teeth/peridontal (Gastrointestinal disorders) | 1 (2)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (4)
Pain::Head/headache (Nervous system disorders) | 3 (4)
Pain::Lymph node (Blood and lymphatic system disorders) | 1 (1)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Pain NOS (General disorders) | 1 (1)
Pain::Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pain::Testicle (Reproductive system and breast disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 6 (23)
Platelets (Blood and lymphatic system disorders) | 6 (37)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (11)
Prolonged QTc interval (Cardiac disorders) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 1 (1)
Pulmonary hypertension (Cardiac disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9 (13)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Secondary Malignancy - possibly related to cancer treatment (Specify, donor cell leukemia) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (2)
Supraventricular and nodal arrhythmia::Sinus bradycardia (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 3 (4)
Thrombotic microangiopathy (e.g., thrombotic thrombocytopenic purpura [TTP] (Vascular disorders) | 1 (1) — or hemolytic uremic syndrome [HUS])
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 4 (9)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 2 (2)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vaginal stenosis/length (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Weight loss (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT00923364/Prot_SAP_000.pdf
  • Informed Consent Form: Recipient Consent (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT00923364/ICF_001.pdf
  • Informed Consent Form: Donor Consent (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT00923364/ICF_002.pdf